CLINICAL TRIAL: NCT04765462
Title: An Open-label, Phase 1/2 Study of Allogeneic γδ T Cell Therapy for the Treatment of Solid Tumors
Brief Title: Allogeneic γδ T Cell Therapy for the Treatment of Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-061
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Malignant Solid Tumours

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic γδ T cell Group (Experimental): Enrolled patients will be administered allogeneic γδ T cells with or without the combinations of traditional therapies, including chemotherapy, targeted therapy, radiotherapy, immune checkpoint inhibitors and others.
  Interventions: Biological: Allogeneic γδ T cells

INTERVENTIONS:
Biological: Allogeneic γδ T cells — Phase 1:Enrolled patents will be administered allogeneic γδ T cells from 2x10^6/kg, 1 x10^7/kg to 5x10^7/kg every 2-4 weeks to determine the recommended dose level.
  Phase 2: Enrolled patents will be administered allogeneic γδ T cells at the recommended dose level to confirm the efficacy.
  Whether or not in combination with other therapies will be determined by research physicians according to the disease status of enrolled patients.

SUMMARY:
The study is to determine the safety, feasibility and efficacy of allogeneic γδ T cell therapy in patients with solid tumors.

DETAILED DESCRIPTION:
This is an open-label, single-center, phase 1/2 study to evaluate the safety, feasibility and efficacy of allogeneic γδ T cell therapy. In phase 1 period, a typical 3+3 dose-escalation design will be used to determine the optimal dose level based on the incidence of dose-limiting toxicity (DLT), which will be recommended as the fixed dose level in the following expansion period and phase 2. The initial infusion dose level will start from 2x10^6/kg to 5x10^7/kg in every 2-4 weeks. Combinations with chemotherapy, targeted therapy, radiotherapy, immune checkpoint inhibitors and other therapies are allowed in this study depending on the disease status of the enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of malignant solid tumors, including patients received surgery, patients with initially diagnosed or pre-treated local advanced/metastatic malignancies, and patients with B-cell non-Hodgkin's lymphomas.
2. Patients should sign informed consent form voluntarily before the trail and comply with the requirements of this study.
3. Age from 18 to 75 years old, gender unlimited.
4. Eastern Cooperative Oncology Group (ECOG) Performance score≤2.
5. Patient with adequate bone marrow reserve (Haemoglobin≥80g/L, Absolute Neutrophil Count (ANC) ≥1×10^6/L, Platelet≥75×10^9/L or ≥50×10^9/L for liver tumors), hepatic function (Aspartate Aminotransferase (AST) / Alanine Aminotransferase (ALT) ≤ 3.0x upper limit of normal or ≤ 5 x ULN for liver tumors or liver metastases, Total bilirubin ≤ 1.5 x ULN), renal function (Creatinine ≤ 1.5 x upper limit of normal (ULN)) and cardiac function (Left ventricular ejection fraction of ≥50% by ECHO).
6. Patient with life expectancy of at least 3 months.
7. Patient without bleeding and coagulation disorders.
8. Patient without obvious genetic diseases.
9. Toxicity from previous antitumor therapy ≤ grade 1 (according to CTCAE version 5.0) or to an acceptable level of inclusion/exclusion criteria (other toxicities such as alopecia and vitiligo considered by the investigator to pose no safety risk to the subject).
10. Male and female patients of reproductive potential must agree to use birth control during the study and for at least 12 weeks post study.

Exclusion Criteria:

1. Patients who received or are to receive any other cell therapy within 4 weeks before the planned day for the first allogeneic γδ T cell administration.
2. Patients who participated or are to participate in other interventional clinical trial within 30 days before the planned day for the first allogeneic γδ T cell administration.
3. Uncontrolled serious active infection (such as sepsis, bacteremia and fungemia, HBV, HCV, HIV, TP, CMV or EBV infection).
4. Systemic steroid therapy or other immune-suppressants (except in cases where the patient is receiving treatment with replacement doses for adrenal insufficiency).
5. Pregnancy or lactation before or during the trial.
6. Patients with history of prior organ or bone marrow transplantation.
7. Patients with systemic vasculitis, or with active or uncontrolled autoimmune diseases, as well as primary or secondary immunodeficiency diseases.
8. History of epilepsy or other active central nervous system disorders.
9. Patients inoculated live vaccine within 6 weeks before screening.
10. Allergic constitution, history of allergies to blood products, known to be allergic to any substances in the protocol(such as Zoledronate or similar).
11. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or any other medical condition that precludes surgery. Also, psychiatric illness/social situations that would limit compliance with study requirements.
12. Any other situations that investigators believe the risk of the subjects is increased or results of the trial are disturbed

Donor Inclusion Criteria:

1. Sign informed consent form.
2. Age 18 years up to the age of 50 (≤50), gender unlimited.
3. Relative to patients (unrestricted to blood relationship).
4. Apheresis available.
5. PLT≥100×109/L with normal APTT or PT.
6. preculture of γδ T cells meets the requirements of massive amplification and detection.

Donor Exclusion Criteria:

1. History of any severe clinical diseases or other severe organic diseases, including any history of clinically significant systematic diseases such as cardiovascular, urinary, circulatory, respiratory, neurological, psychiatric, digestive and endocrine diseases. History of high blood pressure or systolic pressure>140 mmHg, diastolic pressure>90 mmHg in screening stage. Any situation that investigators believe is clinically significant or with other severe diseases unsuitable of apheresis.
2. Arterial thrombosis or venous thrombosis history 12 months prior to the trial or hemorrhagic tendency or history 2 months prior to the trial; oral administration of anticoagulation drugs (e. g. aspirin and warfarin).
3. Active or history of autoimmune diseases including but not restricted to SLE, psoriasis, RA, IBD and HT. Apart from hypothyrosis which can be controlled by hormone replacement therapy, skin diseases without systemic therapy and celiac disease which is fully controlled.
4. HIV-Ab, TP-Ab, HCV-Ab, HBsAg, HBeAg, HBeAb or HBcAb positive.
5. Any symptom, sign or laboratory examination abnormality suggesting acute or subacute infection (e.g. fever, cough, urinary irritation, skin infectious wound).
6. Female who are pregnant or cannot stop lactating.
7. Those who cannot communicate with medical staff due to mental illness or language disabilities.
8. Other unsuitable conditions that investigators believe unsuitable for the donation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) | Baseline to Day 30
  The dose escalation strategy will follow the Food and Drug Administration Guideline for design of early phase clinical trials of cellular therapy products.
Incidence of severe adverse events | Baseline to Day 100
  Safety of the γδ T cell infusion will be based on the risk of treatment-related severe adverse events as identified in the National Cancer Common Terminology Criteria for Adverse Events (CTCAE) version 5.

SECONDARY OUTCOMES:
Objective Response Rate | Baseline to 2years
  Objective clinical response will be assessed by investigators every 2 circles during the treatments and every 2 months after treatment until 2 years after the start of 1st cycle of treatment.
Duration of Response | Baseline to 2years
  The duration of objective response in patients will be recorded until 2years after the start of 1st cycle of treatment
Overall Survival | Baseline to 2years
  Observation for overall survival l (OS) will be recorded until 2years after the start of 1st cycle of treatment.
Progress Free Survival | Baseline to 2years
  Observation for progression-free survival (PFS) will be recorded until 2years after the start of 1st cycle of treatment
Intervention Treatment-related adverse events(AEs) | Baseline to 12 months
  Incidence, nature ,and severity of adverse events will be graded according to the NCI CTCAEv5.0.

OTHER OUTCOMES:
Exploratory research | Baseline to 12 months
  γδ T cells in peripheral blood after infusion will be analysed by TCR or flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, M.D, Principal Investigator — Biotherapeutic Department of Chinese PLA General Hospital; Yanshan Li, Principal Investigator — Biotherapeutic Department of Chinese PLA General Hospital; Kaichao Feng, Principal Investigator — Biotherapeutic Department of Chinese PLA General Hospital
Locations (1):
- Biotherapeutic Department of Chinsese PLA Gereral Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No